CLINICAL TRIAL: NCT05574946
Title: Comparison of Two ACL Reconstruction Techniques: All-inside Versus Complete Tibial Tunnel Technique Using Adjustable Suspensory Fixation
Brief Title: Comparison of Two ACL Reconstruction Techniques: All-inside Versus Complete Tibial Tunnel Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEOALLACL
Record Dates: First submitted 2022-10-06; First posted 2022-10-12 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Anterior Cruciate Ligament Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- All-inside technique (Experimental): Both of the femoral and tibial tunnel will be drilled in a retrograde manner using flip-cutter and femoral and tibial sockets will be created. Graft will be passed from the portal. Adjustable suspensory cortical fixation both on tibial and femoral side will be used.
  Interventions: Procedure: Anterior Cruciate Ligament Reconstruction
- Complete tibial tunnel technique (Active Comparator): Femoral tunnel will be drilled in an inside-outside manner using standard technique. Then the tibial tunnel will be drilled completely. Graft will be passed from the tibial tunnel. Adjustable suspensory cortical fixation both on the tibial and femoral side will be used.
  Interventions: Procedure: Anterior Cruciate Ligament Reconstruction

INTERVENTIONS:
Procedure: Anterior Cruciate Ligament Reconstruction — Anterior Cruciate Ligament Reconstruction with four strand semitendinosus graft

SUMMARY:
This study intends to perform an all-inside and complete tibial tunnel ACL reconstruction technique in 80 patients, and compare the clinical and radiological outcomes of the two surgical procedures through follow-up.

DETAILED DESCRIPTION:
This is a prospective randomized, controlled, single-center clinical trial study on ACL reconstruction surgery technique. In this study, 80 patients with ACL rupture were recruited according to the enrollment criteria. The recruited patients were randomly divided into groups. The ratio of the control group is 1:1. In this study, 40 patients with ACL rupture in the experimental group will be treated with all-inside reconstruction technique, and 40 patients with ACL rupture in the control group will be treated with complete tibial tunnel technique. All operations will be performed with 4-strand autologous semitendinosus tendon. All fixations will be performed using an adjustable cortical suspensory system. After reconstruction, all subjects will participate in the collection of clinical function scores including Marx Activity score, IKDC score, and clinical evaluation including physical examination, joint laxity, CT and MRI imaging analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided informed written written consent;
* Patients aged between 18 and 45;
* Patients undergoing reconstructive surgical treatment of the anterior cruciate ligament (ACL)
* Patients undergoing ACL reconstruction with a 8 mm four-strand semitendinosus autograft

Exclusion Criteria:

* Patients who have not signed informed consent;
* Patients undergoing any additional concomitant ligament repair or reconstruction at the same surgery
* Revision procedures
* Patients unable to lay still in an MRI or CT scanner
* Patients with a torn ACL or previous ACL reconstruction in the contralateral knee.
* Patients who had an excessive tibial slope >12 degrees

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Signal to Noise Quotient | 1 year
  Graft maturation on MRI using T2 Turbo Spin Echo (TSE) sequence without fat saturation

SECONDARY OUTCOMES:
Difference in Computed Tomography (CT) imaging of Tunnels | 1 day, 6 months, 1 year
  Femoral and Tibial Tunnel Morphological Changes
International Knee Documentation Committee (IKDC) | 1 year
  Patient reported outcome measures of symptoms, sports activity & knee function. 0-100 points with 0 (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms)
Marx Activity Rating Score | 1 year
  Clinical Outcomes
Side to side difference in anterior tibial translation | 6 weeks, 3 months, 6 months, 9 months, 1 year
  Anterior tibial translation measured by (Knee laxity Testing device) KT-1000 Arthrometer

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Samsun University, Samsun, Samsun
  - Ahmet E. Okutan, Samsun

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhimani R, Shahriarirad R, Ranjbar K, Erfani A, Ashkani-Esfahani S. Transportal versus all-inside techniques of anterior cruciate ligament reconstruction: a systematic review. J Orthop Surg Res. 2021 Dec 23;16(1):734. doi: 10.1186/s13018-021-02872-x. PMID 34949188
- [Background] Colombet P, Saffarini M, Bouguennec N. Clinical and Functional Outcomes of Anterior Cruciate Ligament Reconstruction at a Minimum of 2 Years Using Adjustable Suspensory Fixation in Both the Femur and Tibia: A Prospective Study. Orthop J Sports Med. 2018 Oct 22;6(10):2325967118804128. doi: 10.1177/2325967118804128. eCollection 2018 Oct. PMID 30364847